CLINICAL TRIAL: NCT07304258
Title: A Prospective, Phase II Clinical Study of HIPEC Combined With NIPS and Tislelizumab Conversion Therapy for Gastric Cancer With Peritoneal Metastasis With Positive Cytology Alone or PCI Score ≤10
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-NIPS-T Trial
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer Peritoneal Metastases
Keywords: HIPEC; NIPS; PD-1
MeSH Terms: interventions — Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel; S 1 (combination); tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental)
  Interventions: Device: HIPEC; Device: NIPS; Drug: Paclitaxel Injection, S-1, tislelizumab

INTERVENTIONS:
Device: HIPEC — HIPEC protocol: Paclitaxel Injection, 75mg/m², D1, D3, D5, for three cycles, followed by a two-week rest before initiating NIPS combined with systemic therapy.
Device: NIPS — Paclitaxel Injection for intraperitoneal perfusion at a dose of 20mg/m² on D1 and D8; Q3W.
Drug: Paclitaxel Injection, S-1, tislelizumab — Paclitaxel Injection: 50mg/m², iv, D1, D8; Q3W; Tegafur Gimeracil Oteracil Potassium Capsules (S-1):For body surface area (BSA) <1.25, 40mg per dose; BSA ≥1.25 to <1.5, 50mg per dose; BSA ≥1.5, 60mg per dose; po, bid, D1-D14; Q3W; Tislelizumab: 200mg per administration, intravenous drip over 30 minutes (not less than 20 minutes and not exceeding 60 minutes), D1, Q3W.

SUMMARY:
This study aims to evaluate the efficacy and safety of HIPEC combined with NIPS and tislelizumab conversion therapy for gastric/gastroesophageal junction cancer with positive cytology alone (CY1P0) or a Peritoneal Carcinomatosis Index (PCI) ≤10

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve patients who have not received chemotherapy, radiotherapy, or any other antitumor therapy prior to the start of the clinical trial;
2. Age between 18 and 75 years;
3. Male or non-pregnant, non-lactating female;
4. Gastric or gastroesophageal junction adenocarcinoma confirmed by gastroscopy and pathological diagnosis;
5. HER-2 negative by immunohistochemistry (IHC), and PD-L1 CPS ≥1;
6. Laparoscopic exploration confirming either positive cytology alone (P0CY1) or peritoneal metastasis (PCI score ≤10);
7. No other distant metastases;
8. Hematological criteria: white blood cell count ≥3.5×10⁹/L, neutrophils ≥1.5×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥90 g/L;
9. Biochemical criteria: ALT ≤2.5×ULN, AST ≤2.5×ULN, total bilirubin ≤1.5×ULN, serum creatinine ≤1.5×ULN;
10. Left ventricular ejection fraction ≥50%;
11. ECOG performance status 0-1;
12. Ability to comply with the study protocol and voluntarily provide signed informed consent.

Exclusion Criteria:

1. Inability to comply with the study protocol or procedures;
2. Known HER2-positive status;
3. Known diagnosis of squamous cell carcinoma, undifferentiated carcinoma, or other histological types of gastric cancer, or adenocarcinoma mixed with other histological types;
4. Current conditions or diseases affecting drug absorption;
5. Patients preoperatively confirmed as unsuitable for conversion therapy;
6. Severe cardiovascular diseases, such as uncontrolled heart failure, coronary artery disease, arrhythmia, or uncontrolled hypertension;
7. Symptomatic active central nervous system metastases (e.g., clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth);
8. Known allergy to the investigational drug(s);
9. Prior treatment with anti-PD-1/PD-L1 antibodies, anti-PD-L2 antibodies, anti-CD137 antibodies, anti-CTLA-4 antibodies, or other drugs/antibodies targeting T-cell co-stimulation or checkpoint pathways;
10. Clinically uncontrolled active infections, such as acute pneumonia, active hepatitis B or C (HBV DNA ≥1×10⁴ copies/mL or >2000 IU/mL despite prior antiviral therapy); Known primary immunodeficiency or active tuberculosis; History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; Known history of human immunodeficiency virus (HIV) infection (HIV antibody positive);
11. Significant malnutrition (weight loss ≥5% within 1 month or >15% within 3 months prior to informed consent, or food intake reduced by ≥50% within 1 week), unless corrected for ≥4 weeks before the first dose of investigational drug;
12. History of other primary malignancies, except:

    * Malignancies in complete remission for at least 2 years prior to enrollment with no required treatment during the study;
    * Adequately treated non-melanoma skin cancer or malignant lentigo with no evidence of recurrence;
    * Adequately treated carcinoma in situ with no evidence of recurrence;
13. Female patients who are pregnant or breastfeeding;
14. Any concomitant illness that, in the investigator's judgment, seriously endangers patient safety or affects study completion;
15. Patients deemed ineligible for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Conversion Rate | The day of surgery
  Proportion of R0 Resection Patients in the ITT Population

SECONDARY OUTCOMES:
1-year PFS rate | 1 year
  Proportion of patients without disease progression or death for at least 1 year from treatment initiation
2-year OS rate | 2 years
  Proportion of patients surviving for at least 2 years from treatment initiation
Progression-free survival（PFS） | 3 years
  Time from enrollment to disease progression or death
Overall survival (OS) | 3 years
Adverse events | 3 years
  Assessment of the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) according to the NCI-CTCAE v5.0 criteria; abnormalities in vital signs and laboratory tests

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Affiliated Hospital of Hebei Medical University, Shijiazhuang, Hebei, China